CLINICAL TRIAL: NCT05995223
Title: Oxygen Uptake Kinetics During Submaximal Exercise in Adults With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Victor Beck, Graduate Research Assistant, University of Nevada, Las Vegas
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: UNLV-2022-489
Record Dates: First submitted 2023-06-29; First posted 2023-08-16 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Down Syndrome
Keywords: Down syndrome; cardiorespiratory fitness; oxygen uptake; cardiac output; mitochondrial oxygen utilization
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Down syndrome (Experimental): Participants will complete a submaximal walking protocol on a motorized treadmill, which consists of 4 times 6 minutes of walking at a moderate intensity speed and incline while their breathing, cardiac output, and muscle oxygen use is measured, with 10 minutes rest in between each bout.
  Interventions: Other: Submaximal exercise protocol
- control without Down syndrome (Experimental): This group of age- and sex-matched participants without Down syndrome will undergo the same testing as participants with Down syndrome
  Interventions: Other: Submaximal exercise protocol

INTERVENTIONS:
Other: Submaximal exercise protocol — Participants will complete a submaximal walking protocol on a motorized treadmill, which consists of 4 times 6 minutes of walking at a moderate intensity speed and incline while their breathing, cardiac output, and muscle oxygen use is measured, with 10 minutes rest in between each bout.

SUMMARY:
This study aims to compare the rate at which oxygen uptake adapts to submaximal, moderate intensity exercise (oxygen uptake kinetics) between adults with and without Down syndrome, to determine the contribution of oxygen uptake kinetics to exercise intolerance of adults with Down syndrome. Additionally, the study will investigate the role of oxygen delivery (by the cardiovascular circuit) and oxygen utilization (in the mitochondria) on the oxygen uptake kinetics of adults with Down syndrome to identify specific areas which adults with Down syndrome could benefit from targeting during exercise training. Overall, this study aims to contribute to the knowledge on the exercise capacity of adults with Down syndrome, in order to improve the way adults with Down syndrome participate in and benefit from exercise.

Participants will perform a maximal exercise test on a treadmill, and walk on a treadmill at a submaximal, moderate intensity speed and incline, during which oxygen uptake at the lungs, cardiac output, and oxygen utilization in the muscle will be measured.

DETAILED DESCRIPTION:
Down syndrome (Ds) is the most common chromosomal disorder, affecting approximately 1 in every 800 live births in the US. In addition to a number of comorbidities, individuals with Ds have low cardiorespiratory fitness. Their low fitness cannot be explained by low levels of physical activity, lack of motivation, or lack of understanding of the test, but rather has a physiological cause. Autonomic dysfunction has been identified as one major contributor to the low cardiorespiratory fitness in individuals with Ds, but it does not fully explain the phenomenon.

Cardiorespiratory fitness is determined by the capacity of the body to produce energy, which largely relies on the ability to take up, deliver, and use oxygen. This process of oxygen transport is governed by the pulmonary, cardiovascular, and muscular system, and the degree to which they work together. At the start of exercise, these three systems respond in a delayed pattern, requiring the body to compensate energy production through anaerobic means, which negatively affect one's exercise tolerance. Thus, the quicker the adaptation of these three systems (i.e. the quicker their kinetics), the better one's ability to perform and tolerate exercise.

The rate of adaption of these oxygen transport system can be quantified by assessing oxygen uptake (pulmonary), cardiac output (cardiovascular), and mitochondrial oxygen utilization (muscle) kinetics, which all show a delayed, exponential increase towards steady state at the start of moderate intensity exercise. The kinetics of these three systems have never been assessed in individuals with Ds, and could provide valuable insights into their low cardiorespiratory fitness and reduced exercise tolerance.

The aim of this research proposal is therefore to determine the differences in kinetics of oxygen uptake, cardiac output, and mitochondrial oxygen utilization between individuals with and without Ds to better understand the underlying physiology and potentially improve healthy by using this knowledge for exercise interventions.

Overall aim: to better understand the relation between oxygen uptake kinetics and cardiorespiratory fitness in individuals with Ds.

Aim 1: To compare the rate of oxygen uptake, cardiac output, and mitochondrial oxygen utilization kinetics in response to submaximal, moderate intensity exercise between adults with and without Ds.

Aim 2: To determine the relation between the rate of oxygen uptake kinetics and the peak oxygen uptake of individuals with Ds.

Determining how oxygen transport affects individuals with Ds during exercise could potentially give more direction into designing exercise sessions and interventions, as their oxygen transport system potentially might need more time to reach the required working level.

General study design. Participants will complete two study visits, during which their cardiorespiratory capacities will be tested using two different treadmill protocols. Familiarization with all study personnel and procedures will take place before actual measurements are performed.

Description data collection visits. Participants will be tested in a postprandial state (>3 h) on 2 separate days (separated by at least 48 hours, but no more than 2 weeks) and will refrain from exercise, alcohol and caffeine for at least 24 h before each study visit. During the first visit, height, weight, and circumferences will be measured. Body composition will be measured using dual energy X-ray absorptiometry (DEXA), and echocardiography will be performed to determined aortic diameter and to screen for any potential residual cardiac deficits common in individuals with Ds. Lastly, participants will perform a graded maximal treadmill exercise test to determine peak oxygen uptake (VO2peak) and to determine the submaximal exercise intensity for the second visit.

The second visit will have participants walk on an intensity associated with 80% of their ventilatory threshold for six minutes while pulmonary oxygen uptake (using breath-by-breath gas exchange analysis), cardiac output (using beat-to-beat blood pressure measurement), and muscle oxygenation (using near-infrared spectroscopy (NIRS)) is measured. This bout of six minutes will be repeated four times, with 10 minutes rest in between. The four bouts will be used to average the three signals, which improves the calculation of kinetic parameters.

Familiarization. Parents/care givers are involved in order to provide a supportive environment for participants and to enhance the parent/caregiver understanding of the research. Prior to study initiation, photographs and video clips of the laboratory and study equipment will be provided to help the participants become comfortable with the laboratory environment and equipment, and the informed consent information is sent to the participants and their parents/care-givers for their review. Familiarization for the participants with Down syndrome will be divided in two parts: they will practice and become accustomed with the treadmill and the equipment for the graded maximal exercise test (very start of the first visit), and they will practice and become accustomed with the procedures for the submaximal exercise protocol (start of the second visit).

ELIGIBILITY:
Inclusion Criteria:

* low active (defined as being involved in less than 30 minutes of moderately-intense physical activity per day);
* diagnosis with Down syndrome trisomy 21 (Down syndrome group only);
* normal thyroid function or stable thyroid function (with medications) for at least 6 months (Down syndrome group only).

Exclusion Criteria:

* asthma or other pulmonary disease;
* severe obesity (defined as BMI >40);
* uncontrolled hypertension (defined as blood pressure >130/80 mmHg);
* congenital heart disease;
* diabetes (defined as Hba1c of >7.5% or use of glucose lowering medication);
* current smoking;
* pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Oxygen uptake kinetics | Through study completion, on average 4 hours
  The finite rate at which oxygen uptake (measured with breath-by-breath gas exchange analysis at the mouth) adapts to a (submaximal) increase in exercise intensity, primarily captured by time constant tau, which describes the time needed to reach 63% of the required, steady state oxygen uptake

SECONDARY OUTCOMES:
Cardiac output kinetics | Through study completion, on average 4 hours
  The finite rate at which cardiac output (calculated from beat-to-beat blood pressure waves) adapts to a (submaximal) increase in exercise intensity, primarily captured by time constant tau, which describes the time needed to reach 63% of the required, steady state cardiac output
Muscle deoxygenation kinetics | Through study completion, on average 4 hours
  The finite rate at which muscle oxygen utilization (measured as the production of deoxyhemoglobin at the muscle) adapts to a (submaximal) increase in exercise intensity, primarily captured by time constant tau, which describes the time needed to reach 63% of the required, steady state muscle oxygen utilization
Steady-state cardiac output | Through study completion, on average 4 hours
  Steady state cardiac output during standing rest and submaximal exercise (in L/min)
Absolute peak oxygen uptake | Through study completion, on average 4 hours
  Peak oxygen uptake (VO2peak; expressed in L/min)
Relative peak oxygen uptake (corrected for total body mass) | Through study completion, on average 4 hours
  Peak oxygen uptake (VO2peak; expressed in ml/kg/min)
Relative peak oxygen uptake (corrected for lean body mass) | Through study completion, on average 4 hours
  Peak oxygen uptake (VO2peak; expressed in L=mL/kg lean body mass/min)
Ventilatory threshold (L/min) | Through study completion, on average 4 hours
  The threshold where ventilation starts to increase at a faster rate than oxygen uptake during a graded maximal exercise test (expressed in L/min)
Ventilatory threshold (%VO2peak) | Through study completion, on average 4 hours
  The threshold where ventilation starts to increase at a faster rate than oxygen uptake during a graded maximal exercise test (expressed as a percentage of VO2peak)
Stroke volume | Through study completion, on average 4 hours
  Stroke volume (mL)
Heart rate | Through study completion, on average 4 hours
  Heart rate (in bpm)
Oxygen uptake efficiency slope | Through study completion, on average 4 hours
  The slope between oxygen uptake (L/min) and the common logarithm of minute ventilation (L/min) during a graded maximal exercise test
Ve/VCO2 slope | Through study completion, on average 4 hours
  The slope between minute ventilation (Ve; L/min) and carbon dioxide production (VCO2; L/min) during a graded maximal exercise test
Lean body mass | Through study completion, on average 4 hours
  Lean body mass determined with Dual Energy X-ray Absorptiometry (DXA) scan in kg

CONTACTS AND LOCATIONS:
Overall Officials: Victor DY Beck, MS, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
De-identified IPD will be made available to other researchers upon request.